CLINICAL TRIAL: NCT04245228
Title: Does a Pre-transplant Health Coaching Intervention for Informal Caregivers of Adult Heart or Lung Transplant Candidates Improve Caregiver-Reported Outcomes?
Brief Title: Wellness Coaching for Caregivers of Thoracic Transplant Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Cassie C. Kennedy, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-008807; R03HL155040 (NIH)
Record Dates: First submitted 2020-01-14; First posted 2020-01-28 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Stress, Psychological; Caregiver Burden
Keywords: Caregiver; Heart Transplant; Lung Transplant; Stress
MeSH Terms: conditions — Stress, Psychological; Caregiver Burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (No Intervention): Routine caregiver transplant education
- Wellness Coaching Intervention (Experimental): Caregivers will be assigned a wellness coach
  Interventions: Behavioral: Wellness Coach

INTERVENTIONS:
Behavioral: Wellness Coach — Trained in motivational interviewing who will call the patient weekly for 12 sessions for an approximately 30-minute intervention
  Arms: Wellness Coaching Intervention

SUMMARY:
Researchers are studying the effects of a health coaching intervention on the stress and burden of caregivers of patients awaiting heart or lung transplant.

DETAILED DESCRIPTION:
This is a randomized trial of health coaching compared to usual care. Caregivers for patients on the adult heart or adult lung transplant waiting list at the Mayo Clinic will undergo informed consent. Consenting participants will be randomized to weekly, 30-minute telephone calls for twelve weeks or usual care. Questionnaires and demographic information will be collected at baseline and after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older who are the primary caregivers of patients listed (active, deferred, or temporarily inactive) for lung, heart/lung, or heart transplantation at Mayo Clinic in Rochester and Jacksonville, FL

Exclusion Criteria:

* Individuals younger than 18 years
* Non-English speaking, non-verbal, or extremely hard of hearing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cassie Kennedy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care Group | Wellness Coaching Intervention
Started (enroll first patients) | 30 | 30
Completed | 30 | 27
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Group | Wellness Coaching Intervention | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (7.2) | 61.9 (7.1) | 62.1 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 16 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 27 | 25 | 52
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 28 | 27 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Perceived Stress Scale (PSS) [Mean (Standard Deviation); unit: units on a scale] — Perceived Stress Scale-10 (PSS-10) is a 10-item tool to evaluate perception of stress during the past month (Cronbach α: 0.74-0.91). The Perceived Stress Scale (PSS) is a self-assessment tool used to measure stress. Individual scores can range from 0 to 40 with higher scores indicating higher perceived stress. Questions are scored 0-4 with scores of 0-13 indicate low; 14-26 indicate moderate; and 27 and above indicate high stress. We will evaluate the PSS of intervention group compared to the change in PSS for the usual care.
  units on a scale | 13.3 (6.5) | 13.4 (7.5) | 13.4 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability
Description: Percentage of participants who completed the study intervention
Time Frame: after completion of the 12-week intervention or between 12-16 weeks after enrollment
Population: Study participants in health coaching or usual care group at the end of study
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Group | Wellness Coaching Intervention
Number analyzed (Participants) | 30 | 30
Participants | 30 | 27

2. Secondary Outcome: Perceived Stress Scale (PSS)
Description: Perceived Stress Scale-10 (PSS-10) is a 10-item tool to evaluate perception of stress during the past month (Cronbach α: 0.74-0.91). The Perceived Stress Scale (PSS) is a self-assessment tool used to measure stress. Individual scores can range from 0 to 40 with higher scores indicating higher perceived stress. Questions are scored 0-4 with scores of 0-13 indicate low; 14-26 indicate moderate; and 27 and above indicate high stress. We will evaluate the PSS of intervention group compared to the change in PSS for the usual care.
Time Frame: after completion of the 12 week intervention or between 12-16 weeks after enrollment.
Population: Post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care Group | Wellness Coaching Intervention
Number analyzed (Participants) | 30 | 27
score on a scale | 14.1 (7.3) | 13.0 (8.2)

ADVERSE EVENTS:
Time Frame: Participants were active in the study for 16 weeks.
Arm/Group | Usual Care Group | Wellness Coaching Intervention
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT04245228/Prot_SAP_000.pdf